CLINICAL TRIAL: NCT01217866
Title: A Retrospective Analysis of a Complete Enseal Laparoscopic Vaginal Assisted Hysterectomy Versus a Traditional Suture Laparoscopic Vaginal Hysterectomy
Brief Title: A Retrospective Review of Enseal Laparoscopic Vaginal Assisted Hysterectomy (LAVH) Versus Traditional LAVH
Status: Completed | Type: Observational
Sponsor: Womens Care (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Principal Investigator, Kathryn OKeeffe MD, MD, Womens Care
Other Study IDs: 1-44206615
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Benign Uterine Disease
Keywords: laparoscopic; vaginal; hysterectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LAVH, techniques: Women aged 35-75 who underwent laparoscopic assisted vaginal hysterectomy via either suture technique vaginally or Enseal coagulation cutting device vaginally
  Interventions: Procedure: Laparoscopic assisted vaginal hysterectomy

INTERVENTIONS:
Procedure: Laparoscopic assisted vaginal hysterectomy — Surgical removal of uterus vaginally

SUMMARY:
Retrospective charts review from one surgeon to compare Group A- cases where the laparoscopic portion of the case used an EN~SEAL device to Group B - the laparoscopic BSO was done using a 3mm EN-SEAL device through 2 lateral 5mm ports.

DETAILED DESCRIPTION:
79 women with benign uterine disease underwent laparoscopic assisted vaginal hysterectomy with or without bilateral salpingo-oophorectomy. Subjects charts were divided into two groups based on surgical technique and the following parameters were reviewed retrospectively: surgical time, blood loss, uterine weight, patient weight, patient age, post operative fever >100.4 F, readmission to hospital within one week, return to operating room within 24 hours, length of hospital stay, and blood transfusion. Group A, N=35 used traditional suture technique vaginally. Group B, N=44 used Enseal coagulation cutting device vaginally.

ELIGIBILITY:
Inclusion Criteria:

* none, observational study

Exclusion Criteria:

* none, observational study

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent Laparoscopically Assisted Vaginal Hysterectomy (LAVH)
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2010-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Surgical time | Operating room time in minutes
  The total time the subject spent in surgery was compared between the two groups
Estimated blood loss | Blood loss during surgery in cc per minute
  The total blood loss in cc per minutes operating was compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Katie O'Keeffe, MD, Principal Investigator — Glens Falls Hospital